CLINICAL TRIAL: NCT06021743
Title: The Role of Immune Semaphorins in Steatotic Liver Disease and Sepsis
Acronym: SepsisFAT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital for Infectious Diseases, Croatia (Other)
Collaborators: Croatian Science Foundation (Other Government)
Responsible Party: Sponsor
Other Study IDs: UHID-08
Record Dates: First submitted 2023-08-27; First posted 2023-09-01 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Steatosis of Liver; Sepsis; Immune Response
MeSH Terms: conditions — Fatty Liver; Sepsis | interventions — Mass Screening

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Sepsis: Patients hospitalized due to the sepsis
  Interventions: Diagnostic Test: Evaluation of the degree of steatosis; Diagnostic Test: Screening for the components of metabolic syndrome; Diagnostic Test: Measurement of serum semaphorin concentrations; Diagnostic Test: Measurement of inflammatory cytokines

INTERVENTIONS:
Diagnostic Test: Evaluation of the degree of steatosis — The degree of steatosis will be estimated using the ultrasound and a method for grading steatosis will be measuring the degree of ultrasound attenuation by hepatic fat using a process based on simultaneous transient elastography (TE) which measures the degree of steatosis.
Diagnostic Test: Screening for the components of metabolic syndrome — Anthropometric measures including height, weight, waist circumference and hip circumference will be measured in all patients. Results of the routine laboratory tests as part of the standard diagnostic procedure will be collected: CRP, leukocyte count, ratio neutrophils and lymphocytes, hemoglobin, platelet count, urea, creatinine, bilirubin, AST, ALT, GGT, ALP, albumins, fasting glucose.
Diagnostic Test: Measurement of serum semaphorin concentrations — Semaphorin concentration will be measured in patient sera by ELISA.
Diagnostic Test: Measurement of inflammatory cytokines — A panel of pro- and anti-inflammatory markers will be determined by flow cytometer microsphere-based assay.

SUMMARY:
The impact of the complex liver immunological network on sepsis outcome is largely unknown. Steatotic liver disease (SLD) is the most common chronic liver disease with prevalence of 25% in European countries. The question remains whether patients with SLD are more prone to bacterial infections and what is the impact of persistent liver inflammation to the systemic response to infection, sepsis course and outcomes. Semaphorins are a large family of secreted and membrane-bound biological response modifiers present in many organ systems that are associated with SLD and development of fibrosis, but also might regulate systemic immune responses in sepsis. This study will investigate the association of semaphorins with sepsis outcomes in patients with SLD.

DETAILED DESCRIPTION:
The liver, with its ability to produce acute phase proteins, complement and cytokines, plays a central role in regulating inflammation. A balanced pro- and anti-inflammatory liver response results in bacterial clearance and resolution of inflammation. Steatotic liver disease (SLD) is the most common chronic liver disease associated with systemic changes in immune response. Although there are numerous immunological links between sepsis and SLD, there is a significant gap in knowledge regarding the role of SLD in sepsis. Semaphorins were recently recognized as one of the key regulators of immune responses; while some suppress immune cells activation, proliferation and production of inflammatory cytokines, others stimulate immune responses. Semaphorins were recently shown to be associated with pathogenesis of viral hepatitis, SLD and progression of fibrosis. However, their role in sepsis is unknown. The hypothesis of this project is that semaphorins are regulators of inflammation in patients with SLD that have impact on sepsis outcome.

ELIGIBILITY:
Inclusion Criteria:

* 2 or more SIRS (Systemic Inflammatory Response Syndrome) criteria (1. Hyperthermia >38.3°C or Hypothermia <36°C; 2. Tachycardia >90 bpm; 3. Tachypnea >20 bpm; 3. Leukocytosis (>12,000 μL-1) or Leukopenia (<4,000 μL-1))
* clinical suspicion of sepsis
* enrolled within 24 hours of hospital admission

Exclusion Criteria:

* no consent
* immunosuppression
* malignancies
* immune diseases
* pregnancy
* HIV infection
* presence of chronic liver disease
* consumption of alcohol > 20 g/day

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients admitted at three clinical departments at UHID that meet inclusion criteria will be offered to participate in the study during a 24-month period.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-02-28 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
Detection of semaphorins in patients with sepsis and SLD | 24 months
  Measurement of semaphorins concentration in serum of patients with SLD and sepsis by enzyme-linked immunosorbent assay (ELISA)
Impact of SLD on sepsis outcomes | 24 months
  Analysis of the impact of SLD and steatosis grade (grade 1 - mild steatosis, 2 - moderate, 3 - severe steatosis) on sepsis complications and outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Neven Papic, MD, PhD, Principal Investigator — School of Medicine, University of Zagreb
Locations (1):
- University Hospital for Infectious Diseases Zagreb, Zagreb, Croatia

IPD SHARING:
Plan to Share IPD: No